CLINICAL TRIAL: NCT05477433
Title: Psychiatric Disorders Related to Diabetes Mellitus Type 1 Among Adolescents in Egypt
Brief Title: Psychiatric Disorders Related to Diabetes Mellitus Type 1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer of neurology and psychiatry,faculty of medicine, Assiut University
Other Study IDs: diabetes mellitus
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus Type 1; Adolescents; Psychiatric Disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: diabetes mellitus type 1 — Pittsburgh Sleep Quality Index "PSQI": It is used to detect sleep disturbance or deficits. The PSQI has a scoring key that can be used to calculate a patient's seven subscores, which range from 0 to 3. The subscores are added together to produce a "global" score that ranges from 0 to 21. A global score of 5 or higher denotes poor sleep quality, The Strengths and Difﬁculties Questionnaire (SDQ) The SDQ is a well-validated screening tool for children and adolescents aged 4-17 years that can identify behavioural and emotional issues,Emotional Avoidance Strategy Inventory for Adolescents (EASI) is used. The EASI-A is a 17-item assessing the use of emotionally avoidant strategies in adolescents and higher scores means significants use avoidant strategies, The Toronto Alexithymia Scale (TAS-20) is a self-administered 20-item questionnaire which assesses difficulties in identifying and describing emotions. TAS scores were significantly higher in alexithymia

SUMMARY:
The most common endocrine illness in children and adolescents is type 1 diabetes. It is distinguished by a lack of insulin synthesis and necessitates daily insulin injections to keep glucose levels under control. As a result, there are numerous medical approaches to its management, such as levels of glycosylated haemoglobin (HbA1c) as a marker of glycemic control during the previous three months and monitoring of blood glucose levels, which affect the patient's mental health and quality of life. Type 1 diabetes complications and poor quality of life are widespread. Diabetes therapy is difficult during puberty and adolescence. Adolescents with T1D have poor metabolic control and a higher rate of acute complications. Because the onset of adolescence is frequently associated with decreased adherence to therapy and an increased risk of psychological illnesses.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females were included.
2. Age ranges from 10 to 19 years.
3. Willing of the parents or the caregivers to participate in the study.
4. Duration of T1DM of at least 1 year.

Exclusion Criteria

1. Adolescents with an intelligence quotient below 70.
2. Adolescents with a history of substance use or psychiatric disorders.
3. Adolescents with medical or other neurological conditions.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be screening for adolescents with diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure frequency of sleep problems with diabetes mellitus type 1 | through study completion, an average of 1 year
Measures frequency of psychiatric problems with diabetes mellitus type 1 | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided